CLINICAL TRIAL: NCT03289715
Title: Evaluation of an On-Demand Humidifier on Neuromuscular Patients Requiring Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ICBE-2-16558
Record Dates: First submitted 2017-09-15; First posted 2017-09-21 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arm 1 (Experimental): on demand humidification
  Interventions: Device: On Demand Humidification system Mark 2

INTERVENTIONS:
Device: On Demand Humidification system Mark 2 — The on demand humidification humidifier is set up to alternate between periods of humidification and no humidification totaling 6 periods of 30 minutes duration each. Thus, the test will consist of 3 cycles of disabled humidification and enabled humidification. Each cycle will be with a different humidification setting to assess which setting is most comfortable. In the second phase, the patient will be treated with the dose they had the best experience with in the first test.

SUMMARY:
Monocenter study to determine and evaluate the optimal amount of humidification doses delivered by the On-Demand humidification system in neuromuscular patients requiring home mechanical ventilation. The patient's perception will be monitored with subjective as well as with objective measurements of the optimum comfortable on-demand humidification doses.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 of age; < 85 years of age
2. Participants with a neuromuscular disorder who:

   1. Require 24 hour mechanical ventilation in some form through tracheostomy, mask or mouth piece
   2. Can be ambulatory for at least a few hours during the day while using a heat and moisture exchange device (HME) or no humidification
   3. Can part of the day use a heated pass-over humidification system while on their ventilator (overnight, for example).
3. Able to provide feedback/articulate via some form of communication
4. Patients using a Trilogy ventilator
5. Invasively ventilated patients that are willing to use a HME device on their way to participate in the study (from home to hospital).
6. Patients that are willing to participate and are able to consent and sign the informed consent form. (Patients with the functional capacity for medical decision-making).

Exclusion Criteria:

1. Clinically unstable, i.e.,

   1. Acute respiratory failure
   2. Participants with refractory hypotension (defined as systolic blood pressure less than 90 mm Hg despite inotropic agents)
   3. Uncontrolled cardiac ischemia or arrhythmias
   4. Any participant determined as inappropriate for the study by the Principal Investigator
2. Patients suffering from metastatic or terminal cancer
3. Patients lacking the functional capacity for medical decision-making.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
optimum comfortable amount of on-demand humidification | 3 hours
  questionnaire based on Borg Scale and Visual Analog scale
optimum comfortable amount of on-demand humidification | 3 hours
  heart rate
optimum comfortable amount of on-demand humidification | 3 hours
  breathing rate
optimum comfortable amount of on-demand humidification | 3 hours
  SpO2
optimum comfortable amount of on-demand humidification | 3 hours
  transcutaneous CO2
optimum comfortable amount of on-demand humidification | 3 hours
  number of mucus clearance events

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No